CLINICAL TRIAL: NCT04051242
Title: XENMATRIX™ AB Surgical Graft for the Repair of Severe Musculotendinous Tissue Damaged by Soft Tissue Trauma
Brief Title: Enhanced Bioscaffold for Volumetric Muscle Loss
Acronym: MTEC-VML
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not complete planned enrollment.
Sponsor: J. Peter Rubin, MD (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, J. Peter Rubin, MD, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19040344
Record Dates: First submitted 2019-06-25; First posted 2019-08-09 (Actual); Results first posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Muscle Loss
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- XenMatrix AB Surgical Graft (Experimental): This study proposes to use XenMatrix™ AB Surgical Graft which has 510(k) approval [#K162193] intended for implantation to reinforce soft tissue where weakness exists and for surgical repair of damaged or ruptured soft tissue. This trial proposes to test the applicability and utility of XenMatrix™ AB Surgical Graft in the restoration of function in the setting of volumetric muscle loss after trauma
  Interventions: Device: XenMatrix™ AB Surgical Graft

INTERVENTIONS:
Device: XenMatrix™ AB Surgical Graft — Graft implantation, radiographic, functional, and electrophysotherapy outcomes will be measured at various time points up to 24-28 weeks post-operatively. A CT scan or MRI will be collected at screening and pre-operative visits to evaluate tissue volume, then again at post-operative Visit 1 and Visit 6. Physical therapy training will be performed as a research procedure following Graft implantation for a maximum of 30 weeks. Additionally, Physical Therapy evaluations will be conducted at screening, pre-op visit 1, post-op, and at post-op Visits 3, and 4. A small core needle biopsy 1-5 grams will be collected at three time points to conduct histomorphological assessment of the tissue prior to Graft implantation (Operative visit, Visit 2 and at Visit 4).

SUMMARY:
This is a prospective, single center study conducted at the University of Pittsburgh designed to test the applicability and utility of XenMatrix™ AB Surgical Graft in the restoration of function in the setting of volumetric muscle loss after soft tissue trauma.

DETAILED DESCRIPTION:
Previously, a human subject clinical trial (NCT01292876, PRO10010500) to evaluate a regenerative medicine approach using ECM for VML treatment was conducted. ECM scaffolds were implanted and combined with aggressive and early physical therapy in 13 subjects, then followed for 24-28 weeks after implantation. Histomorphological assessments collected from core needle biopsies identified formation of new, vascularized, innervated islands of skeletal muscle within the implantation site. Subjects demonstrated increased force production in physical therapy evaluations and improved functional task performance when compared with pre-operative performance. By 6 months after ECM implantation, subjects had a 37.3% improvement in strength and 27.1% improvement in range-of-motion tasks. Additionally, changes in nerve conduction study (NCS) and electromyography (EMG) before and after ECM implantation were measured. 63% of study participants experienced improvements in NCS or EMG within the scaffold remodeling site, indicating clinical improvement in muscle strength. The promising functional and regenerative results from this early study encourages evidence of ECM bioscaffolding as a viable treatment to VML.

This study proposes to use XenMatrix™ AB Surgical Graft which has 510(k) approval [#K162193] intended for implantation to reinforce soft tissue where weakness exists and for surgical repair of damaged or ruptured soft tissue, including abdominal plastic and reconstructive surgery; muscle flap reinforcement; hernia repair including abdominal, inguinal, femoral, diaphragmatic, scrotal, umbilical, and incisional hernias. The graft has an antibiotic coating, specifically, Rifampin and Minocycline. This coating has been shown in preclinical in vitro and in vivo testing to reduce or inhibit microbial colonization on the device. The claim of reduction of bacterial colonization of the device has not yet been established with human clinical data, nor has a clinical impact associated with this claim been demonstrated and will need further investigation. This trial proposes to test the applicability and utility of XenMatrix™ AB Surgical Graft in the restoration of function in the setting of volumetric muscle loss after trauma. 10 subjects will be enrolled for participation in the study. Prior to Graft implantation, subjects will receive a pre-operative course of physical therapy for a maximum time period of 16 weeks. A physical therapist will confirm that functional plateau is reached prior to implantation of the Graft. Following Graft implantation, radiographic, functional, and electrophysotherapy outcomes will be measured at various time points up to 24-28 weeks post-operatively. A CT scan or MRI will be collected at screening and pre-operative visits to evaluate tissue volume, then again at post-operative Visit 1 and Visit 6. Physical therapy training will be performed as a research procedure following Graft implantation for a maximum of 30 weeks. Additionally, Physical Therapy evaluations will be conducted at screening, pre-op visit 1, post-op, and at post-op Visits 3, and 4. A small core needle biopsy 1-5 grams will be collected at three time points to conduct histomorphological assessment of the tissue prior to Graft implantation (Operative visit, Visit 2 and at Visit 4).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 70 years of age and able to provide informed consent
* Civilian, and current or former military personnel are eligible to participate
* Have suffered injury resulting in a structural deficit of a minimum of 20% of the muscle group mass and a functional deficit of a minimum of 25% when compared to a contralateral limb present; or if bilateral injury is present to extremities, the potential surgical extremity is to be compared against normal expected values of a sample population of similar age and gender and evidence of remaining tendon and musculotendinous units that could be surgically repaired with sutures.
* Injuries may encompass a single muscle belly or compartment, whether an area is expected to be repaired by sutures will be determined from imaging studies and physical examination. Muscle groups which originate or attach to the long bones of the extremity, and which directly affect strength and function (i.e., Pectoralis Major, Coracobrachialis, Subscapularis, Teres Major/Minor, Latissimus Dorsi, Supraspinatus, Infraspinatus, Gluteus group, Tensor fasciae latae, Piriformis, and quadratus femoris) will also be included in this clinical trial.
* Have suffered traumatic injury within the last 18 months to the upper and/or lower extremity; Target of 18 months or less but subject's may be enrolled with injury outside this range if the principal investigator determines that there is viable muscle in the injured compartment determined by clinical exam and imaging studies.
* Eligible for study procedures 3 months post injury with stability determined by the Principal Investigator and/ or Physician Co-Investigator
* Willing and able to comply with follow up examinations, radiographic studies, physical therapy, muscle biopsy and laboratory tests.

Exclusion Criteria:

* Inability to provide informed consent
* Poor nutrition (demonstrated by clinically significant abnormal lab results for serum albumin and pre-albumin values, per the investigator's discretion)
* Chronic disease such as congestive heart failure, liver disease, renal disease, or diabetes
* Active and unstable disease state or infection anywhere in the body per Physician's evaluation and determination (demonstrated by stated or medical record history and abnormal lab range for CBC with Differential and Platelet, Liver function and chemistry panel values)
* Known coagulopathy (demonstrated by stated or medical record history of diagnosis)
* Pregnancy (demonstrated by a positive result of a urine pregnancy test)• Diagnosis of cancer within last 12 months and /or actively receiving chemotherapy or radiation treatment
* Subjects with an Axis I diagnosis DSM-IV (e.g., Schizophrenia, Bipolar Disorder). Subjects who are found to be stable on medication and receive psychiatric clearance could be eligible for study participation per the Physician's discretion

  .• Subjects with complete muscle/tendon gaps greater than 5 cm that are obvious on imaging studies and are unlikely to be reasonably repaired with sutures and reinforcement, and will be excluded. The investigators recognize that these findings may not be clear on imaging studies, and that the clinical judgment of the surgeon shall be applied in each case.
* Subjects with a known hypersensitivity to porcine serum products
* Allergies to the antibiotics, Rifampin, minocycline, tetracycline currently associated with the XenMatrix AB Surgical Graft
* Any condition or situation as it relates to the subject's health or safety, that would render concern to the investigators, and therefore preclude subject enrollment in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Peter Rubin, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Aesthetic Plastic Surgery Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dziki J, Badylak S, Yabroudi M, Sicari B, Ambrosio F, Stearns K, Turner N, Wyse A, Boninger ML, Brown EHP, Rubin JP. An acellular biologic scaffold treatment for volumetric muscle loss: results of a 13-patient cohort study. NPJ Regen Med. 2016 Jul 21;1:16008. doi: 10.1038/npjregenmed.2016.8. eCollection 2016. PMID 29302336
- [Background] Han N, Yabroudi MA, Stearns-Reider K, Helkowski W, Sicari BM, Rubin JP, Badylak SF, Boninger ML, Ambrosio F. Electrodiagnostic Evaluation of Individuals Implanted With Extracellular Matrix for the Treatment of Volumetric Muscle Injury: Case Series. Phys Ther. 2016 Apr;96(4):540-9. doi: 10.2522/ptj.20150133. Epub 2015 Nov 12. PMID 26564252

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 subjects were consented, and completed in person screening for the study.
  7 subjects did not meet eligibility criteria. 3 subjects were found to be eligible to proceed to study surgical intervention.
  2 subjects completed the study intervention and received XenMatrix AB. In 1 case, due to a delay from the COVID-19 closure to research at the University of Pittsburgh, the subject no longer met study eligibility, once research was permitted to start.
Period: Overall Study
Arm/Group | XenMatrix AB Surgical Graft
Started | 3
Completed | 1
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: 10 participants were consented and enrolled. Of those three were found to be eligible. One of those was later found to be ineligible, when he was re-evaluated after the University Covid authorization to restart research. Two participants completed the surgical intervention, and one of those completed the final 6 month follow up visit.
Arm/Group | XenMatrix AB Surgical Graft
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] | 38.3 [24 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Extremity Function; as Reported by Participant During a Physical Therapy Evaluation, Pre and Post Study Surgical Intervention, Using the Foot and Ankle Ability Measure (FAAM), Activities of Daily Living (ADL) Subscale Score.
Description: The Foot and Ankle Ability Measure (FAAM) activities of daily living subscale asks respondents to report on whether their activity was limited in the last week due to difficulties with their foot/ankle. The self-assessment uses a 5-point Likert scale from, and has a 6th option, not applicable, if difficulties are not specific to the foot/ankle. Answer choices include No difficulty, slight difficulty, moderate difficulty, extreme difficulty or unable to do. There are two subscales, activities of daily living and sports. For activities of daily living maximum score is 84 and lowest possible score is 0. (For the sports scale the maximum is 28 and the lowest possible score is zero. Higher scores indicate less difficulty with performing the activities. The FAAM sub scores are not totaled together but reported separately). For this subject, due to his injury, the investigators are reporting the Activities of Daily Living Subscale.
Time Frame: Baseline, 6 month follow up
Population: Participant 005 completed the FAAM ADL at baseline, and at 6 months post surgical intervention/implantation of Xenmatrix AB graft.
Measure: Number; unit: score on a scale
Arm/Group | XenMatrix AB Surgical Graft
Number analyzed (Participants) | 1
score on a scale
  Baseline FAAM ADL Sub Score | 69
  6 month follow up FAAM ADL Sub Score | 73

2. Primary Outcome: Extremity Strength in Right and Left Knee (as Measured by Dynamometry Using Newtons, in a Knee Flexion Force Exercise), Pre and Post Surgical Intervention at Baseline and 6 Month Follow up.
Description: Assessment of patient extremity mechanical strength in right and left knee, post implantation of XENMATRIX AB™ Surgical Graft; after skeletal muscle injury as determined by physical therapy assessment using knee flexion force, as measured by dynamometry using newtons. Knee flexion force was measured three times, at each timepoint, so both the mean and lowest and highest score are reported below.
Time Frame: Baseline, 6 month follow up
Population: 005, completed both a presurgical/baseline and post-surgical 6 month follow up analysis.
Measure: Mean (Full Range); unit: Force, units measured in newtons
Arm/Group | XenMatrix AB Surgical Graft
Number analyzed (Participants) | 1
Force, units measured in newtons
  Baseline right knee flexion force | 18.9 [14.5 to 23.6]
  baseline left knee flexion force | 12.2 [9.9 to 13.6]
  6 month right knee flexion force | 191.6 [183.4 to 199.1]
  6 month left knee flexion force | 164.4 [131.4 to 183.4]

3. Secondary Outcome: Number of Participants With Infection With the Use of XENMATRIX AB™ Surgical Graft
Description: Number of Participants with Infection with the Use of XENMATRIX AB™ Surgical Graft. Two participants received the XENMATRIX AB™ Surgical Graft, during their study surgical intervention.
Time Frame: 9-11 months
Measure: Number; unit: participants
Arm/Group | XenMatrix AB Surgical Graft
Number analyzed (Participants) | 2
participants | 0

ADVERSE EVENTS:
Time Frame: Participants were followed after consent/enrollment for up to 11 months. Presurgical activities included screening, eligibility review and a preoperative visit within 30 days of surgical intervention (approximately 3-5 months). After surgical intervention was completed, participants were followed for an additional 6 months, with scheduled follow up visits at 1 month, 3 months, and 6 months post.
Arm/Group | XenMatrix AB Surgical Graft
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XenMatrix AB Surgical Graft (N=2)
parathesia of lower limb (Skin and subcutaneous tissue disorders) | 2 (2)
Pain in left thigh, mid quad (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness, lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
numbness, lower limb (Skin and subcutaneous tissue disorders) | 1 (2)
edema of left ankle (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Please note, there were not enough recruited eligible participants to measure significance. Results are presented from a single enrolled participant who received surgical intervention (graft implantation) on a left calf injury, and completed the 6 month physical therapy evaluation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-02-13): https://cdn.clinicaltrials.gov/large-docs/42/NCT04051242/Prot_SAP_ICF_000.pdf